CLINICAL TRIAL: NCT04477486
Title: Phase 2 Study of the Efficacy and Safety of Venetoclax in Combination With Ibrutinib in Japanese Subjects With Relapsed/Refractory Mantle Cell Lymphoma
Brief Title: Study to Assess Effect of Oral Venetoclax Tablet in Combination With Oral Ibrutinib Capsule on Best Overall Response of Complete Response in Adult Japanese Participants With Relapsed/Refractory Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M20-075
Record Dates: First submitted 2020-07-17; First posted 2020-07-20 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2024-12

CONDITIONS: Mantle Cell Lymphoma (MCL)
Keywords: MCL; Venetoclax; ABT-199; Ibrutinib; Imbruvica
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — ibrutinib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ibrutinib + Venetoclax (Experimental): Participants will receive Ibrutinib Dose A + Venetoclax in various doses until a target dose is reached, for up to 104 weeks, followed by Ibrutinib monotherapy.
  Interventions: Drug: Ibrutinib; Drug: Venetoclax

INTERVENTIONS:
Drug: Ibrutinib — Capsule; Oral
  Other Names: Imbruvica
Drug: Venetoclax — Tablet; Oral
  Other Names: ABT-199; Venclexta; GDC-0199; Venclyxto

SUMMARY:
Mantle Cell Lymphoma (MCL) is a form of Non-Hodgkin Lymphoma (NHL - cancer of the lymphatic system in blood) where cells from outer edge of the lymph nodes, called mantle zone become cancerous. In Japan, MCL accounts for about 3% of all NHL cases. Symptoms of MCL may include enlarged lymph nodes, stomach pain, fever, night sweats, and weight loss. Currently, MCL is not curable with standard therapies. The purpose of this study is to evaluate the safety, efficacy, and effect of venetoclax in combination with ibrutinib on best overall response of complete response in participants with relapsed (return of disease) or refractory (not responding to treatment) (R/R) MCL.

Venetoclax is an investigational drug being developed for the treatment of MCL. Ibrutinib is a drug approved for the treatment of MCL. Participants will receive venetoclax (increasing doses) and ibrutinib (fixed dose) for approximately 104 weeks, followed by ibrutinib alone. Adult participants with R/R MCL will be enrolled. Around 12 participants will be enrolled in Japan.

Participants will receive oral venetoclax tablet and oral ibrutinib capsule for 104 weeks. After 104 weeks, participants will receive ibrutinib once daily until their disease progresses, or they cannot tolerate the medication, or until they do not want to participate in the study.

There may be a higher treatment burden for participants in this study compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, bone marrow biopsies, checking for side effects, and completing questionnaires.

DETAILED DESCRIPTION:
Safety and efficacy data through 09 February 2022 are included in the interim analysis.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed Mantle Cell Lymphoma (MCL) (tumor tissue) by local testing.
* At least 1 measurable site of disease on cross-sectional imaging that is >= 2.0 centimeters (cm) in the longest diameter and measurable in 2 perpendicular dimensions per Computed Tomography (CT).
* At least 1, but no more than 5, prior treatment regimens for MCL including at least 1 prior rituximab/anti-CD20 containing regimen.
* Failure to achieve at least partial response (PR) with, or documented disease progression after, the most recent treatment regimen.

Exclusion Criteria:

* Prior therapy with ibrutinib or other Bruton Tyrosine Kinase (BTK) inhibitors.
* History of other malignancies, except:

  * Malignancy treated with curative intent and with no known active disease present for >= 3 years before the first dose of study drug and felt to be at low risk for recurrence by treating physician.
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  * Adequately treated carcinoma in situ without evidence of disease.
* History or current evidence of central nervous system lymphoma.
* Treatment with any of the following within 7 days prior to the first dose of study drug:

  * Moderate or strong cytochrome P450 3A (CYP3A) inhibitors.
  * Moderate or strong CYP3A inducers.
  * Anticancer therapy, including chemotherapy, radiotherapy, small molecule, and investigational agents, and/or monoclonal antibody <=21 days prior to the first dose of study drug.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2025-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (12):
- Japan (12):
  - NHO Nagoya Medical Center /ID# 221958, Nagoya, Aichi-ken
  - Aichi Cancer Center Hospital /ID# 221565, Nagoya, Aichi-ken
  - Kyushu University Hospital /ID# 223299, Fukuoka, Fukuoka
  - Hokkaido University Hospital /ID# 221662, Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital /ID# 221744, Kobe, Hyōgo
  - National Hospital Organization Mito Medical Center /ID# 224912, Higashi Ibaraki-gun, Ibaraki
  - Ishikawa Prefectural Central Hospital /ID# 224896, Kanazawa, Ishikawa-ken
  - Tohoku University Hospital /ID# 221975, Sendai, Miyagi
  - Duplicate_Okayama University Hospital /ID# 221623, Okayama, Okayama-ken
  - Saitama Medical Center /ID# 224910, Kawagoe-shi, Saitama
  - National Cancer Center Hospital /ID# 221812, Chuo-ku, Tokyo
  - Yamagata University Hospital /ID# 221573, Yamagata, Yamagata

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 13 participants were enrolled across 12 sites in Japan.
Pre-assignment Details: The Full Analysis Set (FAS) included all participants who received at least one dose of study drug and was used for all efficacy analyses (except for those based on IRC assessment), safety, and baseline analyses (N=13). The Per-protocol (PP) population excluded participants with non-evaluable disease at baseline (based on IRC assessment). PP population was used for IRC-assessed endpoints (N=12).
Groups:
- Ibrutinib + Venetoclax: Participants received Ibrutinib 560 mg once daily (QD) + Venetoclax starting at 20 mg QD, gradually ramped up over 5 weeks to a target dose of 400 mg QD. Ibrutinib 560 mg QD + Venetoclax 400 mg QD was continued for up to 104 weeks, followed by 560 mg QD Ibrutinib monotherapy.
Period: Overall Study
Arm/Group | Ibrutinib + Venetoclax
Started | 13
Completed | 0
Not Completed | 13
Not completed — Death | 2
Not completed — Ongoing at Time of Analysis | 11

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (N=13)
Groups:
- Ibrutinib + Venetoclax: Participants received Ibrutinib 560 mg QD + Venetoclax starting at 20 mg QD, gradually ramped up over 5 weeks to a target dose of 400 mg QD. Ibrutinib 560 mg QD + Venetoclax 400 mg QD was continued for up to 104 weeks, followed by Ibrutinib monotherapy.
Arm/Group | Ibrutinib + Venetoclax
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.8 (5.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 13
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Japan | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Best Overall Response of Complete Response (CR), as Assessed by the Independent Review Committee (IRC)
Description: Complete response rate (CRR), defined as the percentage of participants achieving a best overall response of complete response (CR) per the Revised Criteria for Response Assessment for Malignant Lymphoma following the Lugano classification (Cheson 2014), assessed by an Independent Review Committee (IRC).
Time Frame: Week 13
Population: Per-Protocol Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ibrutinib + Venetoclax
Number analyzed (Participants) | 12
percentage of participants | 83.3 [51.6 to 97.9]
Statistical Analysis 1: Comparison: Ibrutinib + Venetoclax; Test type: Superiority — Comparing against a historical reference of 12.5% CRR; p < 0.001, Exact Binomial Distribution

2. Secondary Outcome: Percentage of Participants Achieving Best Overall Response of CR or PR, as Assessed by the IRC
Description: Overall Response Rate (ORR), defined as the percentage of participants with a best overall response of CR or PR, per the Revised Criteria for Response Assessment for Malignant Lymphoma, assessed by an Independent Review Committee (IRC).
Time Frame: Week 104
Reporting Status: Not Posted, anticipated posting 2026-06

3. Secondary Outcome: Percentage of Participants Achieving Best Overall Response of CR as Assessed by the Investigator
Description: Best overall response of CR is defined as the percentage of participants achieving a best overall response of CR for the venetoclax and ibrutinib combination, as assessed by the investigator per the Revised Criteria for Response Assessment for Malignant Lymphoma .
Time Frame: Week 104
Reporting Status: Not Posted, anticipated posting 2026-06

4. Secondary Outcome: Percentage of Participants Achieving Best Overall Response of CR or PR, as Assessed by the Investigator
Description: Best overall response of CR or PR will be evaluated using ORR. The ORR is defined as the percentage of participants with a best overall response of CR or PR, according to the Revised Criteria for Response Assessment for Malignant Lymphoma, as assessed by the investigator.
Time Frame: Week 104
Reporting Status: Not Posted, anticipated posting 2026-06

5. Secondary Outcome: Duration of Response (DOR) for Participants Who Achieved a Best Overall Response of CR or PR, as Assessed by the Investigator
Description: DOR is defined as the time from the first occurrence of response (CR or PR) to disease progression or death, whichever occurs first, according to the Revised Criteria for Response Assessment for Malignant Lymphoma, as assessed by the investigator.
Time Frame: Week 104
Reporting Status: Not Posted, anticipated posting 2026-06

6. Secondary Outcome: DOR for Participants Who Achieved a Best Overall Response of CR or PR, as Assessed by the IRC
Description: DOR is defined as the time from the first occurrence of response (CR or PR) to disease progression or death, whichever occurs first, according to the Revised Criteria for Response Assessment for Malignant Lymphoma, as assessed by the IRC.
Time Frame: Week 104
Reporting Status: Not Posted, anticipated posting 2026-06

7. Secondary Outcome: Undetectable Minimal Residual Disease (uMRD) in Participants Who Achieve a Best Overall Response of CR as Assessed by the Investigator.
Description: MRD rate is defined as the percentage of participants with uMRD who achieve a best overall response of CR, according to the Revised Criteria for Response Assessment for Malignant Lymphoma, as assessed by the investigator.
Time Frame: Week 104
Reporting Status: Not Posted, anticipated posting 2026-06

8. Secondary Outcome: uMRD in Participants Who Achieve a Best Overall Response of CR as Assessed by IRC.
Description: MRD rate is defined as the percentage of participants with uMRD who achieve a best overall response of CR, according to the Revised Criteria for Response Assessment for Malignant Lymphoma, as assessed by the IRC.
Time Frame: Week 104
Reporting Status: Not Posted, anticipated posting 2026-06

9. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from the date of the first dose of study drug (venetoclax or ibrutinib) to the date of investigator-assessed disease progression, using the Revised Response Criteria for Response Assessment for Malignant Lymphoma, or death from any cause, whichever occurs first.
Time Frame: Week 104
Reporting Status: Not Posted, anticipated posting 2026-06

10. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of the first dose of the study drug (venetoclax or ibrutinib) to death from any cause.
Time Frame: Week 104
Reporting Status: Not Posted, anticipated posting 2026-06

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from the start of safety data collection to interim data cut (09 February 2022). Median time participants were followed was 36.1 weeks.
Groups:
- Venetoclax + Ibrutinib: Participants received Ibrutinib 560 mg QD + Venetoclax starting at 20 mg QD, gradually ramped up over 5 weeks to a target dose of 400 mg QD. Ibrutinib 560 mg QD + Venetoclax 400 mg QD was continued for up to 104 weeks, followed by Ibrutinib monotherapy.
Arm/Group | Venetoclax + Ibrutinib
All-Cause Mortality (participants affected / at risk) | 2/13
Serious Adverse Events (participants affected / at risk) | 2/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venetoclax + Ibrutinib (N=13)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
HAEMORRHOIDS (Gastrointestinal disorders) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1)
SQUAMOUS CELL CARCINOMA OF LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venetoclax + Ibrutinib (N=13)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1)
LEUKOPENIA (Blood and lymphatic system disorders) | 4 (7)
NEUTROPENIA (Blood and lymphatic system disorders) | 4 (6)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 3 (5)
ATRIAL FIBRILLATION (Cardiac disorders) | 2 (3)
CARDIAC FAILURE (Cardiac disorders) | 1 (2)
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 1 (1)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1)
CHEILITIS (Gastrointestinal disorders) | 1 (2)
CONSTIPATION (Gastrointestinal disorders) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 7 (8)
NAUSEA (Gastrointestinal disorders) | 3 (6)
STOMATITIS (Gastrointestinal disorders) | 1 (1)
TOOTHACHE (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
GENERALISED OEDEMA (General disorders) | 1 (1)
INJECTION SITE PAIN (General disorders) | 1 (2)
MALAISE (General disorders) | 1 (2)
MUCOSAL INFLAMMATION (General disorders) | 1 (1)
PYREXIA (General disorders) | 1 (1)
HYPERSENSITIVITY (Immune system disorders) | 1 (1)
BODY TINEA (Infections and infestations) | 1 (1)
CANDIDA INFECTION (Infections and infestations) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 1 (2)
HERPES ZOSTER (Infections and infestations) | 1 (1)
IMPETIGO (Infections and infestations) | 1 (1)
LOCALISED INFECTION (Infections and infestations) | 1 (1)
PERIODONTITIS (Infections and infestations) | 1 (1)
PHARYNGITIS (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 2 (2)
SKIN INFECTION (Infections and infestations) | 3 (5)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1)
C-REACTIVE PROTEIN INCREASED (Investigations) | 1 (1)
WEIGHT INCREASED (Investigations) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 3 (5)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (4)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2 (2)
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 (2)
ANOGENITAL WARTS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (2)
DYSGEUSIA (Nervous system disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 2 (2)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PHARYNGEAL ERYTHEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY TRACT OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 (2)
ECZEMA (Skin and subcutaneous tissue disorders) | 1 (1)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 1 (1)
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 1 (2)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 (1)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 (2)
HYPERTENSION (Vascular disorders) | 2 (2)
VASCULAR PAIN (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2023-11-17): https://cdn.clinicaltrials.gov/large-docs/86/NCT04477486/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-16): https://cdn.clinicaltrials.gov/large-docs/86/NCT04477486/SAP_001.pdf